CLINICAL TRIAL: NCT02909530
Title: Comparison Between the Olympus EZ Shot 3Plus 19G and EZ Shot 2 19G in Endoscopic Ultrasound-guided Fine Needle Biopsy of Solid Pancreatic Masses
Brief Title: Comparison Between Olympus EZ Shot 3Plus 19G and EZ Shot 2 19G in EUS-guided FNB of Solid Pancreatic Masses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Alexander Meining, Prof. Dr. Alexander Meining, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 222/16
Record Dates: First submitted 2016-09-07; First posted 2016-09-21 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Pancreatic Neoplasms
Keywords: Endoscopic ultrasound-guided fine needle biopsy; Olympus EZ Shot 3Plus; Olympus EZ Shot 2
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First pass EZ Shot 3Plus then EZ Shot 2 (Active Comparator): Olympus EZ Shot 3Plus will be used to puncture the mass first (Intervention EUS-FNB with EZ Shot 3Plus first), then the 19G and EZ Shot 2 will be used to puncture the pancreatic mass.
  Interventions: Device: EUS-FNB with EZ Shot 3Plus first
- First pass EZ Shot 2 then EZ Shot 3Plus (Active Comparator): Olympus EZ Shot 2 will be used to puncture the mass first (Intervention EUS-FNB with EZ Shot 2 19G first), then the EZ Shot 3Plus will be used to puncture the pancreatic mass.
  Interventions: Device: EUS-FNB with EZ Shot 2 19G first

INTERVENTIONS:
Device: EUS-FNB with EZ Shot 3Plus first — Both needles (EZ Shot 3Plus 19G and EZ Shot 2 19G) will be used for endoscopic ultrasound-guided fine needle biopsy (EUS-FNB) in each patient following a predetermined random order which needle is used to pass through the tumor first.
  Arms: First pass EZ Shot 3Plus then EZ Shot 2
Device: EUS-FNB with EZ Shot 2 19G first — Both needles (EZ Shot 3Plus 19G and EZ Shot 2 19G) will be used for endoscopic ultrasound-guided fine needle biopsy (EUS-FNB) in each patient following a predetermined random order which needle is used to pass through the tumor first.
  Arms: First pass EZ Shot 2 then EZ Shot 3Plus

SUMMARY:
Endoscopic ultrasound-guided fine needle biopsy (EUS-FNB) is a valid and recommended technique for tissue diagnosis of pancreatic masses. However, the diagnostic yield is with a sensitivity of 64%-95% and an accuracy of 78%-94% still very low. The EUS-FNB of pancreatic masses is usually performed with a 22-gauge biopsy needle. The small diameter of the needle is usually responsible for the low yield of tissue samples for histopathological examination. The 19-gauge needles help to overcome the limitations of a 22-gauge needle by acquiring a larger amount of cellular material. Thus, performing EUS-FNB with a 19-gauge needle can maximize tissue acquisition and sample adequacy, which is important for appropriate diagnosis. Contrariwise, the technical success rate for sample retrieval in patients with pancreatic head lesions is significantly lower using the 19-gauge compared to the 22-gauge needle. This is attributable to the technical difficulty to push the needle out of the endoscope in the duodenum. Since about 60% of pancreatic cancers are located in the head region, it is therefore particularly important to improve technical success in these cases. The new 19-gauge biopsy needle "Olympus EZ Shot3 Plus" is more flexible than common biopsy needles such as "EZ Shot2" and should therefore provide improved access to regions like pancreatic head. The aim of this multicenter prospective randomized crossover study is to compare those two needles during EUS-FNB of solid pancreatic masses.

Therefore this study will enroll 40 patients in five German centers with solid pancreatic masses and consecutive indication for EUS-FNB. Both needles will be used in each patient following a predetermined random order.

Primary endpoint is the correct histological diagnosis of the mass assessed by each needle. Technical failure is regarded as a negative histological diagnosis.

Secondary endpoints include a comparison of technical failure using each needle, histological quality, duration of procedure and rate of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* solid pancreatic mass and consecutive indication for EUS-FNB

Exclusion Criteria:

* incapacity to give informed consent
* Haemorrhagic disease, disorder of hemostasis and coagulation (PT <60%, PTT> 42 sec. and platelets <60000/µL)
* oral anticoagulants
* dual antiplatelet therapy with thienopyridines (e.g. clopidogrel)
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Correct histological diagnosis of the mass assessed by each needle | 6 months
  Correct histological diagnosis of the mass assessed by each needle compared to gold standard. Gold standard is primarily positive histology, followed by diagnosis made due to additional methods to assess for malignancy (ultrasound, CT, ERCP, surgically retrieved specimen).

SECONDARY OUTCOMES:
technical failure (inability to push the EUS-FNB needle out the endoscope to perform puncture) | Day one
  Number of failure to push the needle out of the endoscope to perform biopsy counted per needle type.
histological quality of the specimen retrieved (visual analog scale) | 24 months
  Comparison of histological Quality using visual analog scale
histological quality of the specimen retrieved (over all satisfaction) | 24 months
  Comparison of histological Quality using over all satisfaction ("1"<"2", "1"="2", "1">"2")
Duration of procedure | Day one
  time frame between Insertion and extraction of needle or failure to conduct FNB
Adverse events | 24 hours
  Acquisition of immediate adverse events related to the procedure or adverse events in the following 24 hours surveillance period or reported delayed adverse events (over 24 hours) related to the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, Principal Investigator — University Ulm
Locations (4):
- Germany (4):
  - Israelitisches Krankenhaus Hamburg, Hamburg
  - Niel Stensen Kliniken Marienhospital Osnabrück, Osnabrück
  - Klinikum Stuttgart, Katharinenhospital, Stuttgart
  - University Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hann A, Epp S, Veits L, Rosien U, Siegel J, Moschler O, Bohle W, Meining A. Multicenter, randomized comparison of the diagnostic accuracy of 19-gauge stainless steel and nitinol-based needles for endoscopic ultrasound-guided fine-needle biopsy of solid pancreatic masses. United European Gastroenterol J. 2020 Apr;8(3):314-320. doi: 10.1177/2050640619887580. Epub 2019 Nov 7. PMID 32213013